CLINICAL TRIAL: NCT06280560
Title: Impact of Controlled Ovarian Stimulation and Luteal Phase Support on Endometrial Receptivity and Endometrial Senescent Cell Pathological Accumulation: Pilot Study
Brief Title: Impact of IVF Hormonal Therapy on Endometrial Receptivity and Endometrial Senescent Cell Pathological Accumulation
Acronym: HormoSenoRec
Status: Recruiting | Type: Observational
Sponsor: Fundación IVI (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 2109-FIVI-087-FD; PI23/00860 (Other Grant/Funding Number: Instituto de Salud Carlos III, co-funded by European Union)
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Endometrial Receptivity
Keywords: Controled Ovarian Stimulation; Luteal Phase Support; Endometrial Receptivity; Organoid; Senescence; Senolytic; Single Cell Sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Endometrial biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Natural Cycle (NC): No hormonal stimulation
  Interventions: Procedure: Natural Cycle (NC)
- Controlled Ovarian Stimulation (COS) + Luteal Phase Support (LPS): Hormonal fresh transfer protocol
  Interventions: Procedure: Controlled Ovarian Stimulation + Luteal Phase Support
- HRT programmed artificial cycle: Delayed hormonal transfer protocol
  Interventions: Procedure: Hormonal Replacement Therapy programmed artificial cycle
- Endometrial receptivity reference group: No hormonal stimulation
  Interventions: Procedure: Endometrial receptivity reference group

INTERVENTIONS:
Procedure: Controlled Ovarian Stimulation + Luteal Phase Support — Short COS protocol with GnRH antagonist followed by progesterone supplementation. Will be initiated after a negative vaginal ultrasonographic scans to define ovarian quiescence, on days 1 and 2 of the menstrual period. For ovarian stimulation, 150-225 UI /day of FSHrec (GONAL F) will be administered along or in combination with 75 UI/day of HMG (Menopur). From day 6 onwards, HMG/FSHrec will be administered on an individual basis according to the serum E2 levels and transvaginal ovarian ultrasound scans and GnRH antagonist (Orgalutran) 0.25 mg /day is introduced as soon as a follicle of 14 mms diameter has achieved. hCGrec (6500 IU, Ovitrelle) will be administered when 7 or 8 follicles with a maximum diameter of >17-18 mms will observed. 400 mg of micronized vaginal progesterone will be administered (200 mg twice a day vaginal route), during 5 days. An endometrial biopsy and a blood sample will be obtained 7 days after hCG administration (hCH+7)
  Groups: Controlled Ovarian Stimulation (COS) + Luteal Phase Support (LPS)
Procedure: Hormonal Replacement Therapy programmed artificial cycle — 6 mg of oestradiol orally administered starting the first day of the menstrual period, followed by an endometrial scan 10-days later, and when a 7 mms triple line endometrium has seen by vaginal ultrasound scan, 800 mg of micronized vaginal progesterone (400 mg twice a day vaginal route), during five days, will be added to the oestrogen therapy. An endometrial biopsy and a blood sample will be obtained on day 5 of progesterone administration (P+5)
  Groups: HRT programmed artificial cycle
Procedure: Natural Cycle (NC) — No hormonal stimulation. From day 6 of the menstrual period, follicular growth will be evaluated. As soon as a follicle reaches 17mm in diameter, ovulation test strips will be provided to assess LH levels in the first morning urine. The participant will report the positive and will be scheduled for sampling seven days later. An endometrial biopsy and a blood sample will be obtained 7 days after LH peak (LH+7)
  Groups: Natural Cycle (NC)
Procedure: Endometrial receptivity reference group — Recruited among women belonging to the oocyte donation program and will follow the procedures described above for the Natural Cycle group. No hormonal stimulation. From day 6 of the menstrual period, follicular growth will be evaluated. As soon as a follicle reaches 17mm in diameter, ovulation test strips will be provided to assess LH levels in the first morning urine. The participant will report the positive and will be scheduled for sampling seven days later. An endometrial biopsy and a blood sample will be obtained 7 days after LH peak (LH+7)
  Groups: Endometrial receptivity reference group

SUMMARY:
Both controlled ovarian stimulation (COS) and frozen embryo transfer has become an integral part of in vitro fertilization (IVF) treatment. Fresh embryo transfer is usually performed by providing Luteal Phase Support (LPS) with progesterone after COS. Frozen embryo transfer (FET) is usually performed in artificial cycles with hormone replacement treatment (HRT), in which exogenous progesterone is administered, although it can also be performed in a Natural Cycle (without hormone supplementation) (NC). There is evidence that the supraphysiologic levels of estradiol and progesterone during COS+LPS and HRT could lead to morphologic and biochemical endometrial modifications, altering endometrial receptivity and lowering implantation and pregnancy rates.

We hypothesize that the supraphysiologic hormone levels required for both COS+LPS, and HRT may be inducing alterations in endometrial composition and function, specifically the chronic accumulation of senescent cells; either due to an excessive hormonal induction, a lack of clearance due to a deficit of uNKs, or a combination of both, ultimately affecting both endometrial receptivity and decidualization, worsening IVF outcomes.

The in vitro clearance of endometrial senescent cells by selective induction of apoptosis has been found to enhance the decidualization capacity of the rest of Endometrial Stromal Cells (EnSC), which could represent in a future adjuvant strategy to reduce the potentially deleterious effects of supraphysiologic hormone levels and improve reproductive outcomes in IVF patients.

The results derived from this project would have a direct impact on clinical practice. First, the results would allow us to evaluate, based on experimental data, potential endometrial side effects of stimulation protocols commonly used in IVF treatments. In addition, in the case of finding a pathological accumulation of senescent cells affecting endometrial receptivity, we will be able to in vitro evaluate the effectiveness of adjuvant senolytic (drugs designed to specifically remove senescent cells) compounds to in vitro improve the expression of endometrial receptivity markers, as a first step to demonstrate the effectiveness of their use in improving the reproductive outcomes of IVF patients.

ELIGIBILITY:
Study group (subfertile IVF patients).

* Inclusion Criteria: Women aged 18-45 years, BMI ≥ 18.5- 30.
* Exclusion criteria: Women presenting any uterine disease that affects the endometrial cavity, or with a thin or irregular endometrium, altered karyotypes, thrombophilias, or uncorrected systemic or endocrine diseases will be excluded.

Endometrial receptivity reference group (oocyte donors).

* Inclusion criteria: women aged between 18 and 35 years, BMI ≥ 18.5- 25.
* Exclusion criteria: Any cases of DIU presence, hormonal contraceptives at least during the last three months, altered karyotypes, thrombophilias, or uncorrected systemic or endocrine diseases will be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist in 45 women undergoing IVF treatment for fertility problems and who, as indicated by their clinical practice, will be subjected to one of the following hormonal protocols (fifteen participants per group) (Natural Cycle, Controled Ovarian Stimulation + Luteal Phase Support, Hormone Replacement Therapy).
  Additionally, as an endometrial receptivity reference group, we will recruit a population of 15 women with proven fertility belonging to the oocyte donation program in an endometrial cycle without hormonal stimulation (natural cycle).
  The 60 participants will be recruited at the IVI-RMA Valencia clinic (Valencia).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Endometrial receptivity | through study completion, an average of 2 years
  To evaluate in vitro (on cells) endometrial receptivity markers such as prolactin, Prolactin, IGFBP1, FOXO1, HOXA-10, CLU, SCAS5, DIO, VEGF, TGFβ, CD34, CD31, CD44, MMPs, IL-15, IL-11, IL-6, LIF, Glycodelin, β-catenin, ALCAM, IGF-1R, c-KIT, SMAD3, etc

SECONDARY OUTCOMES:
Senescent Cell Pathological Accumulation | through study completion, an average of 2 years
  To evaluate in vitro (on cells) the presence of senescence markers such as lipofuscin granules (SentraGor or Sudan Black B), NF-kB, p-16, p-21, p38, P-p38, p53, cGAS, STRING, γH2AX, carbonyl proteins, etc

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Domínguez Hernández, PhD, Principal Investigator — IVI Foundation, Valencia, Valencia, Spain
Locations (1):
- IVI-RMA Valencia Clinic, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
Anonymized results from Single Cell Sequencing will be uploaded to public databases belonging to Gene Expression Omnibus-NCBI for free access by researchers.

REFERENCES:
- [Background] Aplin JD, Stevens A. Use of 'omics for endometrial timing: the cycle moves on. Hum Reprod. 2022 Apr 1;37(4):644-650. doi: 10.1093/humrep/deac022. PMID 35147196
- [Background] Birch J, Gil J. Senescence and the SASP: many therapeutic avenues. Genes Dev. 2020 Dec 1;34(23-24):1565-1576. doi: 10.1101/gad.343129.120. PMID 33262144
- [Background] Boretto M, Cox B, Noben M, Hendriks N, Fassbender A, Roose H, Amant F, Timmerman D, Tomassetti C, Vanhie A, Meuleman C, Ferrante M, Vankelecom H. Development of organoids from mouse and human endometrium showing endometrial epithelium physiology and long-term expandability. Development. 2017 May 15;144(10):1775-1786. doi: 10.1242/dev.148478. Epub 2017 Apr 25. PMID 28442471
- [Background] Boretto M, Maenhoudt N, Luo X, Hennes A, Boeckx B, Bui B, Heremans R, Perneel L, Kobayashi H, Van Zundert I, Brems H, Cox B, Ferrante M, Uji-I H, Koh KP, D'Hooghe T, Vanhie A, Vergote I, Meuleman C, Tomassetti C, Lambrechts D, Vriens J, Timmerman D, Vankelecom H. Patient-derived organoids from endometrial disease capture clinical heterogeneity and are amenable to drug screening. Nat Cell Biol. 2019 Aug;21(8):1041-1051. doi: 10.1038/s41556-019-0360-z. Epub 2019 Aug 1. PMID 31371824
- [Background] Bourgain C, Devroey P. The endometrium in stimulated cycles for IVF. Hum Reprod Update. 2003 Nov-Dec;9(6):515-22. doi: 10.1093/humupd/dmg045. PMID 14714588
- [Background] Brighton PJ, Maruyama Y, Fishwick K, Vrljicak P, Tewary S, Fujihara R, Muter J, Lucas ES, Yamada T, Woods L, Lucciola R, Hou Lee Y, Takeda S, Ott S, Hemberger M, Quenby S, Brosens JJ. Clearance of senescent decidual cells by uterine natural killer cells in cycling human endometrium. Elife. 2017 Dec 11;6:e31274. doi: 10.7554/eLife.31274. PMID 29227245
- [Background] Burton GJ, Jauniaux E, Charnock-Jones DS. Human early placental development: potential roles of the endometrial glands. Placenta. 2007 Apr;28 Suppl A:S64-9. doi: 10.1016/j.placenta.2007.01.007. Epub 2007 Mar 8. PMID 17349689
- [Background] Burton GJ, Redman CW, Roberts JM, Moffett A. Pre-eclampsia: pathophysiology and clinical implications. BMJ. 2019 Jul 15;366:l2381. doi: 10.1136/bmj.l2381. PMID 31307997
- [Background] Check JH, Wilson C, Choe JK, Amui J, Brasile D. Evidence that high serum progesterone (P) levels on day of human chorionic gonadotropin (hCG) injection have no adverse effect on the embryo itself as determined by pregnancy outcome following embryo transfer using donated eggs. Clin Exp Obstet Gynecol. 2010;37(3):179-80. PMID 21077517
- [Background] Cindrova-Davies T, Fogarty NME, Jones CJP, Kingdom J, Burton GJ. Evidence of oxidative stress-induced senescence in mature, post-mature and pathological human placentas. Placenta. 2018 Aug;68:15-22. doi: 10.1016/j.placenta.2018.06.307. Epub 2018 Jun 19. PMID 30055665
- [Background] Clevers H. Modeling Development and Disease with Organoids. Cell. 2016 Jun 16;165(7):1586-1597. doi: 10.1016/j.cell.2016.05.082. PMID 27315476
- [Background] Cox LS, Redman C. The role of cellular senescence in ageing of the placenta. Placenta. 2017 Apr;52:139-145. doi: 10.1016/j.placenta.2017.01.116. Epub 2017 Jan 16. PMID 28131318
- [Background] Deane JA, Cousins FL, Gargett CE. Endometrial organoids: in vitro models for endometrial research and personalized medicine. Biol Reprod. 2017 Jan 1;97(6):781-783. doi: 10.1093/biolre/iox139. No abstract available. PMID 29106468
- [Background] Deryabin P, Griukova A, Nikolsky N, Borodkina A. The link between endometrial stromal cell senescence and decidualization in female fertility: the art of balance. Cell Mol Life Sci. 2020 Apr;77(7):1357-1370. doi: 10.1007/s00018-019-03374-0. Epub 2019 Nov 15. PMID 31728580
- [Background] Deryabin PI, Borodkina AV. Stromal cell senescence contributes to impaired endometrial decidualization and defective interaction with trophoblast cells. Hum Reprod. 2022 Jun 30;37(7):1505-1524. doi: 10.1093/humrep/deac112. PMID 35604371
- [Background] Devroey P, Bourgain C, Macklon NS, Fauser BC. Reproductive biology and IVF: ovarian stimulation and endometrial receptivity. Trends Endocrinol Metab. 2004 Mar;15(2):84-90. doi: 10.1016/j.tem.2004.01.009. PMID 15036255
- [Background] Dominguez F, Avila S, Cervero A, Martin J, Pellicer A, Castrillo JL, Simon C. A combined approach for gene discovery identifies insulin-like growth factor-binding protein-related protein 1 as a new gene implicated in human endometrial receptivity. J Clin Endocrinol Metab. 2003 Apr;88(4):1849-57. doi: 10.1210/jc.2002-020724. PMID 12679483
- [Background] Dominguez F, Gadea B, Mercader A, Esteban FJ, Pellicer A, Simon C. Embryologic outcome and secretome profile of implanted blastocysts obtained after coculture in human endometrial epithelial cells versus the sequential system. Fertil Steril. 2010 Feb;93(3):774-782.e1. doi: 10.1016/j.fertnstert.2008.10.019. Epub 2008 Dec 4. PMID 19062008
- [Background] Evans GE, Phillipson GTM, Sykes PH, McNoe LA, Print CG, Evans JJ. Does the endometrial gene expression of fertile women vary within and between cycles? Hum Reprod. 2018 Mar 1;33(3):452-463. doi: 10.1093/humrep/dex385. PMID 29370409
- [Background] Evans J, Hannan NJ, Edgell TA, Vollenhoven BJ, Lutjen PJ, Osianlis T, Salamonsen LA, Rombauts LJ. Fresh versus frozen embryo transfer: backing clinical decisions with scientific and clinical evidence. Hum Reprod Update. 2014 Nov-Dec;20(6):808-21. doi: 10.1093/humupd/dmu027. Epub 2014 Jun 10. PMID 24916455
- [Background] Frances-Herrero E, Juarez-Barber E, Campo H, Lopez-Martinez S, de Miguel-Gomez L, Faus A, Pellicer A, Ferrero H, Cervello I. Improved Models of Human Endometrial Organoids Based on Hydrogels from Decellularized Endometrium. J Pers Med. 2021 Jun 3;11(6):504. doi: 10.3390/jpm11060504. PMID 34205034
- [Background] Garcia-Alonso L, Handfield LF, Roberts K, Nikolakopoulou K, Fernando RC, Gardner L, Woodhams B, Arutyunyan A, Polanski K, Hoo R, Sancho-Serra C, Li T, Kwakwa K, Tuck E, Lorenzi V, Massalha H, Prete M, Kleshchevnikov V, Tarkowska A, Porter T, Mazzeo CI, van Dongen S, Dabrowska M, Vaskivskyi V, Mahbubani KT, Park JE, Jimenez-Linan M, Campos L, Kiselev VY, Lindskog C, Ayuk P, Prigmore E, Stratton MR, Saeb-Parsy K, Moffett A, Moore L, Bayraktar OA, Teichmann SA, Turco MY, Vento-Tormo R. Mapping the temporal and spatial dynamics of the human endometrium in vivo and in vitro. Nat Genet. 2021 Dec;53(12):1698-1711. doi: 10.1038/s41588-021-00972-2. Epub 2021 Dec 2. PMID 34857954
- [Background] Groothuis PG, Dassen HH, Romano A, Punyadeera C. Estrogen and the endometrium: lessons learned from gene expression profiling in rodents and human. Hum Reprod Update. 2007 Jul-Aug;13(4):405-17. doi: 10.1093/humupd/dmm009. PMID 17584823
- [Background] Haouzi D, Assou S, Mahmoud K, Tondeur S, Reme T, Hedon B, De Vos J, Hamamah S. Gene expression profile of human endometrial receptivity: comparison between natural and stimulated cycles for the same patients. Hum Reprod. 2009 Jun;24(6):1436-45. doi: 10.1093/humrep/dep039. Epub 2009 Feb 26. PMID 19246470
- [Background] Hernandez-Segura A, Nehme J, Demaria M. Hallmarks of Cellular Senescence. Trends Cell Biol. 2018 Jun;28(6):436-453. doi: 10.1016/j.tcb.2018.02.001. Epub 2018 Feb 21. PMID 29477613
- [Background] Horcajadas JA, Minguez P, Dopazo J, Esteban FJ, Dominguez F, Giudice LC, Pellicer A, Simon C. Controlled ovarian stimulation induces a functional genomic delay of the endometrium with potential clinical implications. J Clin Endocrinol Metab. 2008 Nov;93(11):4500-10. doi: 10.1210/jc.2008-0588. Epub 2008 Aug 12. PMID 18697870
- [Background] Horcajadas JA, Riesewijk A, Polman J, van Os R, Pellicer A, Mosselman S, Simon C. Effect of controlled ovarian hyperstimulation in IVF on endometrial gene expression profiles. Mol Hum Reprod. 2005 Mar;11(3):195-205. doi: 10.1093/molehr/gah150. Epub 2005 Feb 4. PMID 15695772
- [Background] Huang R, Fang C, Xu S, Yi Y, Liang X. Premature progesterone rise negatively correlated with live birth rate in IVF cycles with GnRH agonist: an analysis of 2,566 cycles. Fertil Steril. 2012 Sep;98(3):664-670.e2. doi: 10.1016/j.fertnstert.2012.05.024. Epub 2012 Jun 15. PMID 22704632
- [Background] Ishihara O, Araki R, Kuwahara A, Itakura A, Saito H, Adamson GD. Impact of frozen-thawed single-blastocyst transfer on maternal and neonatal outcome: an analysis of 277,042 single-embryo transfer cycles from 2008 to 2010 in Japan. Fertil Steril. 2014 Jan;101(1):128-33. doi: 10.1016/j.fertnstert.2013.09.025. Epub 2013 Oct 23. PMID 24268706
- [Background] Jin J, Richardson L, Sheller-Miller S, Zhong N, Menon R. Oxidative stress induces p38MAPK-dependent senescence in the feto-maternal interface cells. Placenta. 2018 Jul;67:15-23. doi: 10.1016/j.placenta.2018.05.008. Epub 2018 May 17. PMID 29941169
- [Background] Junovich G, Mayer Y, Azpiroz A, Daher S, Iglesias A, Zylverstein C, Gentile T, Pasqualini S, Markert UR, Gutierrez G. Ovarian stimulation affects the levels of regulatory endometrial NK cells and angiogenic cytokine VEGF. Am J Reprod Immunol. 2011 Feb;65(2):146-53. doi: 10.1111/j.1600-0897.2010.00892.x. PMID 20618181
- [Background] Kilicdag EB, Haydardedeoglu B, Cok T, Hacivelioglu SO, Bagis T. Premature progesterone elevation impairs implantation and live birth rates in GnRH-agonist IVF/ICSI cycles. Arch Gynecol Obstet. 2010 Apr;281(4):747-52. doi: 10.1007/s00404-009-1248-0. Epub 2009 Oct 28. PMID 19862542
- [Background] Kolibianakis E, Bourgain C, Albano C, Osmanagaoglu K, Smitz J, Van Steirteghem A, Devroey P. Effect of ovarian stimulation with recombinant follicle-stimulating hormone, gonadotropin releasing hormone antagonists, and human chorionic gonadotropin on endometrial maturation on the day of oocyte pick-up. Fertil Steril. 2002 Nov;78(5):1025-9. doi: 10.1016/s0015-0282(02)03323-x. PMID 12413988
- [Background] Kusama K, Yamauchi N, Yoshida K, Azumi M, Yoshie M, Tamura K. Senolytic treatment modulates decidualization in human endometrial stromal cells. Biochem Biophys Res Commun. 2021 Sep 24;571:174-180. doi: 10.1016/j.bbrc.2021.07.075. Epub 2021 Jul 27. PMID 34330061
- [Background] Labarta E, Martinez-Conejero JA, Alama P, Horcajadas JA, Pellicer A, Simon C, Bosch E. Endometrial receptivity is affected in women with high circulating progesterone levels at the end of the follicular phase: a functional genomics analysis. Hum Reprod. 2011 Jul;26(7):1813-25. doi: 10.1093/humrep/der126. Epub 2011 May 2. PMID 21540246
- [Background] Lancaster MA, Knoblich JA. Organogenesis in a dish: modeling development and disease using organoid technologies. Science. 2014 Jul 18;345(6194):1247125. doi: 10.1126/science.1247125. Epub 2014 Jul 17. PMID 25035496
- [Background] Libby VR, Wilson R, Kresak A, Cameron C, Redline R, Mesiano S, Weinerman R. Superovulation with gonadotropin-releasing hormone agonist or chorionic gonadotropin for ovulation trigger differentially affects leukocyte populations in the peri-implantation mouse uterus. F S Sci. 2021 May;2(2):198-206. doi: 10.1016/j.xfss.2021.03.003. Epub 2021 Mar 20. PMID 35559753
- [Background] Lucas ES, Vrljicak P, Muter J, Diniz-da-Costa MM, Brighton PJ, Kong CS, Lipecki J, Fishwick KJ, Odendaal J, Ewington LJ, Quenby S, Ott S, Brosens JJ. Recurrent pregnancy loss is associated with a pro-senescent decidual response during the peri-implantation window. Commun Biol. 2020 Jan 21;3(1):37. doi: 10.1038/s42003-020-0763-1. PMID 31965050
- [Background] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Background] Martinez-Conejero JA, Simon C, Pellicer A, Horcajadas JA. Is ovarian stimulation detrimental to the endometrium? Reprod Biomed Online. 2007 Jul;15(1):45-50. doi: 10.1016/s1472-6483(10)60690-6. PMID 17623534
- [Background] Maru Y, Tanaka N, Itami M, Hippo Y. Efficient use of patient-derived organoids as a preclinical model for gynecologic tumors. Gynecol Oncol. 2019 Jul;154(1):189-198. doi: 10.1016/j.ygyno.2019.05.005. Epub 2019 May 14. PMID 31101504
- [Background] McLernon DJ, Maheshwari A, Lee AJ, Bhattacharya S. Cumulative live birth rates after one or more complete cycles of IVF: a population-based study of linked cycle data from 178,898 women. Hum Reprod. 2016 Mar;31(3):572-81. doi: 10.1093/humrep/dev336. Epub 2016 Jan 18. PMID 26783243
- [Background] Melo MA, Meseguer M, Garrido N, Bosch E, Pellicer A, Remohi J. The significance of premature luteinization in an oocyte-donation programme. Hum Reprod. 2006 Jun;21(6):1503-7. doi: 10.1093/humrep/dei474. Epub 2006 Apr 28. PMID 16648153
- [Background] Menon R, Boldogh I, Hawkins HK, Woodson M, Polettini J, Syed TA, Fortunato SJ, Saade GR, Papaconstantinou J, Taylor RN. Histological evidence of oxidative stress and premature senescence in preterm premature rupture of the human fetal membranes recapitulated in vitro. Am J Pathol. 2014 Jun;184(6):1740-51. doi: 10.1016/j.ajpath.2014.02.011. Epub 2014 May 12. PMID 24832021
- [Background] Montenegro IS, Kuhl CP, Schneider RA, Zachia SA, Durli ICLO, Terraciano PB, Rivero RC, Passos EP. Use of clomiphene citrate protocol for controlled ovarian stimulation impairs endometrial maturity. JBRA Assist Reprod. 2021 Feb 2;25(1):90-96. doi: 10.5935/1518-0557.20200056. PMID 33118715
- [Background] Montoya-Botero P, Polyzos NP. The endometrium during and after ovarian hyperstimulation and the role of segmentation of infertility treatment. Best Pract Res Clin Endocrinol Metab. 2019 Feb;33(1):61-75. doi: 10.1016/j.beem.2018.09.003. Epub 2018 Sep 13. PMID 30770200
- [Background] Nikas G, Develioglu OH, Toner JP, Jones HW Jr. Endometrial pinopodes indicate a shift in the window of receptivity in IVF cycles. Hum Reprod. 1999 Mar;14(3):787-92. doi: 10.1093/humrep/14.3.787. PMID 10221715
- [Background] Roque M, Haahr T, Geber S, Esteves SC, Humaidan P. Fresh versus elective frozen embryo transfer in IVF/ICSI cycles: a systematic review and meta-analysis of reproductive outcomes. Hum Reprod Update. 2019 Jan 1;25(1):2-14. doi: 10.1093/humupd/dmy033. PMID 30388233
- [Background] Roque M, Lattes K, Serra S, Sola I, Geber S, Carreras R, Checa MA. Fresh embryo transfer versus frozen embryo transfer in in vitro fertilization cycles: a systematic review and meta-analysis. Fertil Steril. 2013 Jan;99(1):156-162. doi: 10.1016/j.fertnstert.2012.09.003. Epub 2012 Oct 3. PMID 23040524
- [Background] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Evidence of impaired endometrial receptivity after ovarian stimulation for in vitro fertilization: a prospective randomized trial comparing fresh and frozen-thawed embryo transfer in normal responders. Fertil Steril. 2011 Aug;96(2):344-8. doi: 10.1016/j.fertnstert.2011.05.050. Epub 2011 Jul 6. PMID 21737072
- [Background] Simon C, Mercader A, Garcia-Velasco J, Nikas G, Moreno C, Remohi J, Pellicer A. Coculture of human embryos with autologous human endometrial epithelial cells in patients with implantation failure. J Clin Endocrinol Metab. 1999 Aug;84(8):2638-46. doi: 10.1210/jcem.84.8.5873. PMID 10443653
- [Background] Suhorutshenko M, Kukushkina V, Velthut-Meikas A, Altmae S, Peters M, Magi R, Krjutskov K, Koel M, Codoner FM, Martinez-Blanch JF, Vilella F, Simon C, Salumets A, Laisk T. Endometrial receptivity revisited: endometrial transcriptome adjusted for tissue cellular heterogeneity. Hum Reprod. 2018 Nov 1;33(11):2074-2086. doi: 10.1093/humrep/dey301. PMID 30295736
- [Background] Turco MY, Gardner L, Hughes J, Cindrova-Davies T, Gomez MJ, Farrell L, Hollinshead M, Marsh SGE, Brosens JJ, Critchley HO, Simons BD, Hemberger M, Koo BK, Moffett A, Burton GJ. Long-term, hormone-responsive organoid cultures of human endometrium in a chemically defined medium. Nat Cell Biol. 2017 May;19(5):568-577. doi: 10.1038/ncb3516. Epub 2017 Apr 10. PMID 28394884
- [Background] Unfer V, Casini ML, Gerli S, Costabile L, Mignosa M, Di Renzo GC. Phytoestrogens may improve the pregnancy rate in in vitro fertilization-embryo transfer cycles: a prospective, controlled, randomized trial. Fertil Steril. 2004 Dec;82(6):1509-13. doi: 10.1016/j.fertnstert.2004.07.934. PMID 15589851
- [Background] Venetis CA, Kolibianakis EM, Papanikolaou E, Bontis J, Devroey P, Tarlatzis BC. Is progesterone elevation on the day of human chorionic gonadotrophin administration associated with the probability of pregnancy in in vitro fertilization? A systematic review and meta-analysis. Hum Reprod Update. 2007 Jul-Aug;13(4):343-55. doi: 10.1093/humupd/dmm007. Epub 2007 Apr 3. PMID 17405832
- [Background] Wang W, Vilella F, Alama P, Moreno I, Mignardi M, Isakova A, Pan W, Simon C, Quake SR. Single-cell transcriptomic atlas of the human endometrium during the menstrual cycle. Nat Med. 2020 Oct;26(10):1644-1653. doi: 10.1038/s41591-020-1040-z. Epub 2020 Sep 14. PMID 32929266
- [Background] Yousefzadeh MJ, Zhu Y, McGowan SJ, Angelini L, Fuhrmann-Stroissnigg H, Xu M, Ling YY, Melos KI, Pirtskhalava T, Inman CL, McGuckian C, Wade EA, Kato JI, Grassi D, Wentworth M, Burd CE, Arriaga EA, Ladiges WL, Tchkonia T, Kirkland JL, Robbins PD, Niedernhofer LJ. Fisetin is a senotherapeutic that extends health and lifespan. EBioMedicine. 2018 Oct;36:18-28. doi: 10.1016/j.ebiom.2018.09.015. Epub 2018 Sep 29. PMID 30279143
- [Background] Zhao Y, Garcia J, Kolp L, Cheadle C, Rodriguez A, Vlahos NF. The impact of luteal phase support on gene expression of extracellular matrix protein and adhesion molecules in the human endometrium during the window of implantation following controlled ovarian stimulation with a GnRH antagonist protocol. Fertil Steril. 2010 Nov;94(6):2264-71. doi: 10.1016/j.fertnstert.2010.01.068. Epub 2010 Mar 12. PMID 20226447
- [Background] Zhu X, Niu Z, Ye Y, Xia L, Chen Q, Feng Y. Endometrium cytokine profiles are altered following ovarian stimulation but almost not in subsequent hormone replacement cycles. Cytokine. 2019 Feb;114:6-10. doi: 10.1016/j.cyto.2018.11.002. Epub 2018 Dec 20. PMID 30562675
- [Background] Lozano-Torres B, Estepa-Fernández A, Rovira M, Orzáez M, Serrano M, Martínez-Máñez R, Sancenón F. The chemistry of senescence. Nat Rev Chem. 2019;3:426-441. doi: 10.1038/s41570-019-0108-0.
- [Background] Organization WH. Infertility prevalence estimates 1990-2021. 2023.